CLINICAL TRIAL: NCT05780034
Title: A Phase I Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Malignancy Activity of AC676 in Patients With Relapsed/Refractory B-cell Malignancies
Brief Title: A Study of AC676 for the Treatment of Relapsed/Refractory B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC676-001
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory B-cell Malignancies
Keywords: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Mantle Cell Lymphoma (MCL); Follicular Lymphoma (FL); Non-Germinal Center B-cell (Non-GCB) Diffuse Large B-cell Lymphoma (DLBCL); Marginal Zone Lymphoma (MZL; Waldenström Macroglobulinemia (WM); Non-Hodgkin Lymphoma (NHL); Bruton's tyrosine kinase-BTK; BTK Degrader; AC676; AC0676
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AC676 Dose Escalation (Experimental): Participants will receive an assigned dose of AC676 in a 28-days cycle.
  Interventions: Drug: AC676

INTERVENTIONS:
Drug: AC676 — AC676 will be given orally (PO) on a 28-day cycle.

SUMMARY:
This clinical trial is evaluating a drug called AC676 in participants with Relapsed/Refractory B-cell Malignancies. The main goals of the study are to:

* Identify the recommended dose of AC676 that can be given safely to participants
* Evaluate the safety profile of AC676
* Evaluate the pharmacokinetics of AC676
* Evaluate the effectiveness of AC676

DETAILED DESCRIPTION:
AC676-001 is a Phase I, first-in-human, open-label, multi-center dose-escalation study of AC676 given as a single agent. AC676 is an investigational medicinal product that is an orally bioavailable BTK degrader for the treatment of B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients, at least 18 years-of-age at the time of signature of the informed consent form (ICF).
2. Patients with histologically confirmed relapsed/refractory Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL), Mantle Cell Lymphoma (MCL), Follicular Lymphoma (FL), non-GCB Diffuse Large B-cell Lymphoma (DLBCL), Marginal Zone Lymphoma (MZL), or Waldenström Macroglobulinemia (WM).
3. Must have received at least 2 prior systemic therapies or have no other therapies to provide significant clinical benefit in the opinion of the Investigator or who are not amenable (intolerability, patient choice) to standard therapies.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Treatment with any of the following:

   * Small molecule anti-cancer drugs within 5 half-lives or 2 days (whichever is longer, not to exceed 14 days).
   * Systemic chemotherapy within 14 days.
   * Radiation therapy within 14 days
   * Biologics (Antibodies) treatment within 28 days,
   * Radioimmunoconjugates or toxin conjugates within 12 weeks.
   * Prior Chimeric antigen receptor (CAR) T cell therapy (and prior use of immunoglobulin replacement therapy to treat associated adverse events) within 3 months. For patients with DLBCL, no prior CAR- T therapy is allowed.
   * Autologous or allogenic stem cell transplant within 100 days and must not have ongoing graft-versus-host disease (GVHD) and no ongoing therapy to treat GVHD.
2. History of central nervous system lymphoma/leukemia in remission for less than 2 years.
3. Medical history of active bleeding within 2 months prior to study entry, or susceptible to bleeding by the judgement of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) from AC676 monotherapy | From cycle 1 day 1 to Cycle 1 day 28. Cycles are 28 days.
Incidence of treatment-emergent adverse events (TEAEs) and clinically significant Grade 3 or higher laboratory abnormalities using CTCAE v5.0 criteria. | Approximately 18 months
Maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) | Approximately 18 months

SECONDARY OUTCOMES:
Pharmacokinetic Analysis: area under the plasma concentration-time curve over the dosing interval (AUC(0-inf)) | Up to approximately 20 weeks
Pharmacokinetic Analysis: area under the plasma concentration-time curve from over the dosing interval (AUC(0-tau)) | Up to approximately 20 weeks
Pharmacokinetic Analysis: maximum plasma concentration (Cmax) | Up to approximately 20 weeks
Pharmacokinetic Analysis: time to maximum plasma concentration (tmax) | Up to approximately 20 weeks
Pharmacokinetic Analysis: terminal elimination half-life (t1/2) | Up to approximately 20 weeks
Objective Response Rate (ORR) in patients receiving AC676 | Approximately 18 months
Duration of Response (DOR) in patients receiving AC676 | Approximately 18 months
Time to Response (TTR) in patients receiving AC676 | Approximately 18 months
Disease Control Rate (DCR) in patients receiving AC676 | Approximately 18 months
Progression Free Survival rate (PFS) in patients receiving AC676 | Approximately 18 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No